CLINICAL TRIAL: NCT06737601
Title: ESWT vs Orthosis in Trigger Finger Treatment: Prospective Randomized Clinical Study
Brief Title: ESWT vs Orthosis in Trigger Finger
Acronym: SWinTF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWinTF
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2024-12

CONDITIONS: Trigger Finger
Keywords: extracorporeal shock waves therapy; trigger finger; orthesis; conservative treatment
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: PROSPECTIVE RANDOMIZED CLINICAL TRIAL
Who Masked: Investigator
Masking Description: Given the nature of the therapy, it is not possible to blind the operators or patients. The medical staff responsible for collecting the disease scores, however, will be blind regarding the assignment of patients to one or the other group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESWT group (Experimental): 3 shock waves sessions, weekly, EDF 1500 pulses, 0.01-0,05 mJ/mm2 (minilith Storz, Swiss)
  Interventions: Device: shock waves
- orthesis group (No Intervention): use of metacarpophalangeal orthosis for 4-6 weeks

INTERVENTIONS:
Device: shock waves — three sessions, weekly frequency
  Arms: ESWT group

SUMMARY:
Recently, two works have proposed the application of Extracorporeal Shock Waves Therapy (ESWT) in the treatment of trigger finger. Yildirim and colleagues (2016) compared shock waves with corticosteroid infiltration. both methods proved effective at 6 months. The authors suggested that shock wave treatment could be a valid non-invasive therapy option for this pathology. Chen and colleagues (2021) analyzed two different shock wave protocols [high and low Energy Density Flux (EDF)] vs placebo. All treatment groups showed improvements within 6 months. The high-energy treatment (EDF 0.01 mj/mm2) demonstrated greater effects on clinical remission and functional recovery compared to the other two groups in the study. The aim of our study is to compare the effects of shock waves vs the use of the orthosis.

DETAILED DESCRIPTION:
Trigger finger, also called flexor digitorum stenosing tenosynovitis, is a pathological condition characterized by a size discrepancy between the flexor tendon/tendon sheath and the A1 pulley, located in the metacarpal head. This pathology causes pain and blockage of the flexion tendon of the finger, with a frequency of 2.6% in the general population, with a higher incidence in the female population, especially in the fifth and sixth decade. The 4th, 3rd and 1st fingers are most involved. trigger finger limits daily activities, such as grasping and holding objects with handles, manipulating coins and buttoning.

The diagnosis is based on the clinical history of transient locking of the finger when flexed with subsequent painful snapping when extended. The trigger phenomenon can be preceded by pain and joint stiffness. The instrumental study, with ultrasound and/or MRI, allows you to monitor the severity of the disease, identify the underlying cause and decide on the appropriate treatment. Surgical treatment should be reserved for those who do not respond to conservative treatment and desire definitive resolution.

A consensus was conducted to identify the consensus treatment guideline for trigger finger, including nonsteroidal anti-inflammatories, orthoses, corticosteroid infiltration and percutaneous release, and surgery. No evidence was found to support the use of nonsteroidal anti-inflammatory drugs. There has been evidence regarding the use of an orthosis, because by immobilizing the finger joint, it would prevent the occurrence of a trigger. Corticosteroid infiltration was effective, albeit with shorter-term effects than the orthosis, with high rates of relapses and exacerbations after 6 months. Surgical treatment is reserved for those who do not benefit from conservative therapy and need a definitive result.

ELIGIBILITY:
Inclusion Criteria:

* Grade 2~3 trigger finger according to Quinnell classification
* problem that has been occurring for at least 3 months

Exclusion Criteria:

* Previous treatment via physiotherapy, local corticosteroid injection or surgical release for trigger finger within 3 months prior to recruitment.

  * Presence of musculoskeletal disease or previous nerve injury to the upper extremities.
  * Multiple trigger finger.
  * contraindications to treatment with ESWT: local infection; epilepsy; malignant tumor; inflammatory arthritis; cardiac arrhythmia or cardiac pacemaker; and pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
recovery of pain | From enrollment to 1, 3 and 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Trigger frequency | From enrollment to 1, 3 and 6 months
  A 0 to 10-point trigger finger rating scale to evaluate this parameter according to a previous study (Tarbhai et al., 2012). This scale is also used to evaluate the severity of the trigger (ST) and the functional impact of the trigger (FIT).
Quick-Disabilities of the Arm, Shoulder, and Hand (QuickDASH) | From enrollment to 1, 3 and 6 months
  The QuickDASH measures the effect of finger problems on function in terms of pain and disability. The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Solarino, M.D., Study Director — University of Bari

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Quinnell RC. Conservative management of trigger finger. Practitioner. 1980 Feb;224(1340):187-90. No abstract available. PMID 7367373
- [Background] Tarbhai K, Hannah S, von Schroeder HP. Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am. 2012 Feb;37(2):243-9, 249.e1. doi: 10.1016/j.jhsa.2011.10.038. Epub 2011 Dec 20. PMID 22189188
- [Background] Chen YP, Lin CY, Kuo YJ, Lee OK. Extracorporeal Shockwave Therapy in the Treatment of Trigger Finger: A Randomized Controlled Study. Arch Phys Med Rehabil. 2021 Nov;102(11):2083-2090.e1. doi: 10.1016/j.apmr.2021.04.015. Epub 2021 May 21. PMID 34029555
- [Background] Yildirim P, Gultekin A, Yildirim A, Karahan AY, Tok F. Extracorporeal shock wave therapy versus corticosteroid injection in the treatment of trigger finger: a randomized controlled study. J Hand Surg Eur Vol. 2016 Nov;41(9):977-983. doi: 10.1177/1753193415622733. Epub 2016 Sep 28. PMID 26763271
- [Background] Huisstede BM, Hoogvliet P, Coert JH, Friden J; European HANDGUIDE Group. Multidisciplinary consensus guideline for managing trigger finger: results from the European HANDGUIDE Study. Phys Ther. 2014 Oct;94(10):1421-33. doi: 10.2522/ptj.20130135. Epub 2014 May 8. PMID 24810861
- [Background] Bianchi S, Gitto S, Draghi F. Ultrasound Features of Trigger Finger: Review of the Literature. J Ultrasound Med. 2019 Dec;38(12):3141-3154. doi: 10.1002/jum.15025. Epub 2019 May 20. PMID 31106876
- [Background] Makkouk AH, Oetgen ME, Swigart CR, Dodds SD. Trigger finger: etiology, evaluation, and treatment. Curr Rev Musculoskelet Med. 2008 Jun;1(2):92-6. doi: 10.1007/s12178-007-9012-1. PMID 19468879
- [Background] Akhtar S, Bradley MJ, Quinton DN, Burke FD. Management and referral for trigger finger/thumb. BMJ. 2005 Jul 2;331(7507):30-3. doi: 10.1136/bmj.331.7507.30. No abstract available. PMID 15994689
- See also: Related Info — https://sitod.it/